CLINICAL TRIAL: NCT02516553
Title: An Open Label, Phase Ia/Ib Dose Finding Study With BI 894999 Orally Administered Once a Day in Patients With Advanced Malignancies, With Repeated Administration in Patients With Clinical Benefit
Brief Title: BI 894999 First in Human Dose Finding Study in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1367.1; 2015-001111-12 (EudraCT Number)
Record Dates: First submitted 2015-07-27; First posted 2015-08-06 (Estimated); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Neoplasms; NUT Carcinoma
Keywords: NUT midline carcinoma
MeSH Terms: conditions — Neoplasms | interventions — BI 894999

ARMS (22):
- Phase Ia - Schedule A: 0.2 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule A: 0.5 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule A: 1 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule A: 1.5 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule A: 2 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule A: 5 mg BI 894999 (Experimental): Once daily continuous oral intake in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 1.5 mg BI 894999 (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 2 mg BI 894999 (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 2.5 mg BI 894999 (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule C: 5/2.5 mg BI 894999 (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule C: 6/3 mg BI 894999 (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule C: 7/3.5 mg BI 894999 (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL patients) (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999
- Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL patients) (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999
- Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ib - Schedule B: 2.5 mg BI 894999 (NC patients) (Experimental): Once daily intermittent oral intake with two weeks on treatment followed by one week off in 3-week cycles.
  Interventions: Drug: BI 894999
- Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC patients) (Experimental): Once daily loading dose on Day 1 followed by six days daily intake of maintenance dose, followed by one week off, repeated every two weeks in cycles of 28 days.
  Interventions: Drug: BI 894999

INTERVENTIONS:
Drug: BI 894999 — film-coated tablets

SUMMARY:
This study is open to adults with different types of advanced cancer (solid tumours). The study is also open to patients with diffuse large B-cell lymphoma in whom previous treatment was not successful. In some countries, adolescents who are at least 15 years old and who are diagnosed with NUT carcinoma can also participate. No standard treatment exists for this rare and aggressive form of cancer.

The purpose of this study is to find out the highest dose of BI 894999 that people can tolerate.

BI 894999 is tested for the first time in humans. Participants take tablets once daily. The study also tests whether participants can tolerate BI 894999 better when taken continuously or with breaks in between.

Participants can stay in the study as long as they benefit from the treatment and can tolerate it.

The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

For all patients

* Age 18 years or older at the time of signature of the informed consent.
* Life expectancy of at least 12 weeks after the start of the treatment according to the investigator's judgement
* Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. For women of childbearing potential using a contraceptive pill, an additional barrier method is necessary due to the potential CYP3A4 inducing effect of BI894999. Male patients having a partner of childbearing potential must use condoms and ensure their partner is using a highly effective method of birth control as described above, during the trial and for at least three months after the end of the trial * Any female who has experienced menarche and does not meet the criteria for "women not of childbearing potential" as described below.

Women not of childbearing potential are defined as: women who are postmenopausal (12 months with no menses without an alternative medical cause) or who are permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

- Written informed consent consistent with ICH-GCP and local legislation

For patients with solid tumours

* Patients with a histologically or cytologically confirmed diagnosis of an advanced unresectable and/or metastatic, malignant solid tumour, who have failed conventional treatment or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies
* Age ≥ legal age to be adult for the given country at the time of signature of the informed consent. For NC patients, age 15 years or older at the time of signature of the informed consent ( in Germany and South Korea, only legally adult patients may be included
* Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score 0 or 1 at the time of screening. A score of 2 is allowed for NUT carcinoma patients
* Recovery of therapy-related toxicities from previous chemotherapy, tyrosine kinase inhibitors, hormone therapy, immunotherapy, antibodies, vaccine therapy, or radiotherapy to CTCAE ≤ grade 1 (with the exception of alopecia, peripheral sensory neuropathy grade 2)
* Life expectancy of at least 12 weeks after the start of the treatment according to the investigator's judgement
* Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. For women of childbearing potential using a contraceptive pill, an additional barrier method is necessary due to the potential CYP3A4 inducing effect of BI894999. Male patients having a partner of childbearing potential must use condoms and ensure their partner is using a highly effective method of birth control as described above, during the trial and for at least three months after the end of the trial treatment
* Written informed consent consistent with ICH-GCP and local legislation. For adolescent NC patients aged 15 years to < legal adult age, written assent of the patient and written informed consent of the parents (both or one according to national regulation) or legal guardian of the adolescent
* Written informed consent for tumour biopsies in the escalation phase Ia

  * Optional for those patients until extension of the MTD cohort,
  * Optional for the patients in the extension of MTD cohort at the same time points as described below for the expansion phase. For these patients in the extension of the MTD cohort, if they have an accessible lesion for biopsy, they will be offered optional consent for tumour biopsies
* In addition, all patients included in the expansion Phase Ib must:
* Have been diagnosed with one of the four types of tumours selected:

  * small cell lung cancer (SCLC)
  * metastatic castrate resistant prostate cancer (mCRPC)
  * colorectal cancer (CRC)
  * NUT carcinoma (NC) (for which the "midline" origin is not a prerequisite)
* Have failed conventional treatments or who are not amenable to standard therapies (per criterion 1) that specifically include for:

  * SCLC: a platinum-based therapy (previous treatment with topotecan is not mandatory)
  * mCRPC: a hormonal agent (abiraterone, enzalutamide, or apalutamide) and a taxane (docetaxel or cabazitaxel)
  * CRC: fluoropyrimidine, oxaliplatin and irinotecan, bevacizumab for patients eligible to this treatment and an anti-epidermal growth factor receptor (EGFR) in RAS (Rat Sarcoma Virus) wild type metastatic CRC.
* Have measurable disease (radiated lesions and lesions used for biopsy do not qualify as target lesions), according to RECIST 1.1 (R09-0262) (for NC patients only nonmeasurable disease is acceptable); or according to PCWG3 (R17-3377) for the mCRPC cohort (see point 5 of inclusion criteria below, specific to mCRPC patients)
* Have progressive disease within the last 6 months, according to RECIST 1.1 (R09-0262) or according to PCWG3 (R17-3377) for the mCRPC cohort (see point 5 of inclusion criteria below, specific to mCRPC patients). NC patients do not need to show progression per RECIST 1.1 (for example, if newly diagnosed).
* Have a tumour lesion accessible for biopsies (pre- and at steady state under treatment in Cycle 1, ideally from the same anatomic lesion) (except for mCRPC patients having only bone metastases or for patients with therapeutic INR because of treatment with a vitamin K antagonist or a novel oral anticoagulant. Biopsies are optional for NC patients
* Give written informed consent for two tumour biopsies, one at screening and one after start of treatment, between Day 8 and Day 11 of Cycle 1 (or between day 3 and day 8 if the day of biopsy in Cycle 1 needs to be moved as explained in Section 3.1) (when applicable)
* In addition, all patients in the mCRPC expansion cohort of Phase Ib must have:
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Radiographic evidence of metastatic prostate cancer (stage M1 or D2). Distant metastases evaluable by bone scan, CT scan, or MRI within 28 days before the start of study treatment.
* PSA ≥ 5 ng/mL (if no measurable disease by RECIST 1.1)
* Prior surgical or chemical castration with a serum testosterone of <50 ng/dL (< 1.7 nmol/L) by luteinizing hormone releasing level hormone (LHRH) agonist or antagonist, or by abiraterone or by enzalutamide or apalutamide. If the actual method of castration is LHRH agonist or antagonist, the patient must be willing to continue the use of LHRH agonist or antagonist during protocol treatment.
* Progressive disease defined as at least one of the following:

  * Progressive measurable disease: using conventional solid tumour criteria RECIST 1.1
  * Bone scan progression: at least two new lesions on bone scan plus a rising PSA as described in point c below
  * Increasing PSA level: at least two consecutive rising PSA values over a reference value (PSA no.1) taken at least 1 week apart. A third PSA (PSA no. 3) is required to be > than PSA no. 2; if not, a fourth PSA (PSA no. 4) is required to be > to PSA no. 2

In patients with DLBCL

* Patients with histologically confirmed DLBCL who have failed 2 or more lines of systemic therapy including an anti-CD-20 therapy and an anthracycline or who are not amenable to standard therapies but have an indication for therapy as per investigator's judgement. Standard therapies may also include but are not limited to CAR-T cells therapy, depending on approved therapies in the country where the patient is treated
* ECOG Performance Status 0, 1 or 2 at the time of screening
* Measurable disease (radiated lesions do not qualify as target lesions) according to according to RECIL 2017 on the CT scan part of the FDG/PET-CT scan
* Recovery of therapy-related toxicities from previous anti-lymphoma therapy to CTCAE <= grade 1 (with the exception of alopecia, peripheral sensory neuropathy grade 2)
* written informed consent for tumour biopsies (optional)
* Further inclusion criteria apply

Exclusion criteria:

For all patients:

* Inability to swallow tablets
* Additional other serious illness, concomitant non-oncological disease (e.g. active infectious disease including an active infection with SARS-CoV-2 confirmed by a PCR test or had one in the prior 6 weeks or active hepatitis (Hep) B infection as defined by positive Hep B DNA test, active Hep C infection as defined by positive Hep C RNA test and human immunodeficiency virus (HIV) infection (positive result in established HIV diagnostic assay), or ongoing toxicity from prior therapies considered by the investigator to potentially compromise patient's safety in this trial
* Serum creatinine greater than 1.5 mg/dL (>132 µmol/L, SI unit equivalent)
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Treatment with other investigational drugs or participation in another clinical interventional trial within the past four weeks or within five times the half-life of the previous investigational drug, whichever is shorter, before start of therapy or concomitant with this trial
* Patients unable to comply with the protocol
* Patients who are actively abusing alcohol or drugs. Since no alcohol or drug testing is required per protocol, it is at the investigator's discretion to determine abuse.

For patients with solid tumours:

* Additional other serious illness , concomitant non-oncological disease (e.g. active infectious disease or known chronic Hepatitis B/Hepatitis C infection and HIV), or ongoing toxicity from prior therapies considered by the investigator to potentially compromise patient's safety in this trial
* History or presence of cardiovascular abnormalities deemed clinically relevant by the investigator such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to study entry.Left Ventricular Ejection Fraction (LVEF) less than 50% at baseline
* Clinical evidence of symptomatic progressive brain or leptomeningeal disease during the last 28 days before the start of treatment with BI 894999
* Absolute neutrophil count less than 1500/mm^3
* Platelet count less than 100 000/mm^3
* Bilirubin greater than 1.5 mg/dL (>26 µmol/L, SI unit equivalent) (except known Gilbert's syndrome, accepted up to 2 mg/dL or up to 34.2 µmol/L in this case)
* Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases, greater than five times the upper limit of normal)
* Treatment with other investigational drugs or participation in another clinical interventional trial within the past four weeks (past two weeks for NC patients) or within five times the half-life of the previous investigational drug, whichever is the shorter, before start of therapy or concomitant with this trial
* Systemic anti-cancer therapy within four weeks (past two weeks for NC patients) or five times the half-life of the drug, whichever is shorter. Radiotherapy given for curative intent or other than palliative radiotherapy within the past four weeks before start of therapy or concomitantly with this trial. This These restrictions does not apply to LHRH agonists or antagonists, steroids (given at a stable dose in the last four weeks) used for palliative intent, bisphosphonates, and denosumab and to palliative radiotherapy (no wash out required)

For patients with DLBCL:

* Patient is eligible for curative salvage high dose therapy followed by stem cell transplant.
* Primary central nervous system (CNS) lymphoma or known CNS involvement
* Prior allogeneic bone marrow or stem cell transplant
* High-dose therapy with stem cell support <3 months prior to visit 1
* AST or ALT >2.5 x upper limit of normal (CTCAE grade 2 or higher)
* Total bilirubin >1.5 x upper limit of normal (CTCAE grade 2 or higher)
* Absolute neutrophil count <1.0 x 10^9/L(without growth factor support)
* Platelets <100 x 10^9/L (without transfusions)
* Significant concurrent medical disease or condition which according to the investigator's judgement would either compromise patient safety or interfere with the evaluation of the safety of the test drug, e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry, cardiac arrhythmia requiring therapy with the exception of extra systoles or minor conduction abnormalities
* Chronic or ongoing infection requiring treatment at the time of enrolment or within the previous two weeks, e.g. active infectious disease or known Hepatitis B/Hepatitis C infection, HIV
* Systemic anti-DLBCL therapy within the past two weeks or five times the half-life of the drug, whichever is shorter (palliative radiotherapy and agents used for palliative reasons for example steroids and bisphosphonates, are allowed)
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - Brussels - HOSP Jules Bordet, Anderlecht
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
- France (4):
  - HOP Timone, Marseille
  - HOP Hôtel-Dieu, Nantes
  - HOP Saint-Louis, Paris
  - INS Gustave Roussy, Villejuif
- Universitätsklinikum Tübingen, Tübingen, Germany
- Samsung Medical Center, Seoul, South Korea
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Schoffski P, Machiels JP, Rottey S, Sadrolhefazi B, Musa H, Marzin K, Awada A. Phase Ia dose-escalation trial with the BET protein inhibitor BI 894999 in patients with advanced or metastatic solid tumours. Eur J Cancer. 2023 Sep;191:112987. doi: 10.1016/j.ejca.2023.112987. Epub 2023 Jul 11. PMID 37556913
- See also: Related Info — https://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, Phase Ia/Ib dose finding study with BI 894999 orally administered once a day in patients with advanced malignancies with repeated administration in patients with clinical benefit.
Pre-assignment Details: For Phase Ib - Schedule B SCLC, Phase Ib - Schedule B mCRPC, DMC decided on 28Nov2018 to lower the dose of SCLC and mCRPC due to safety concern, thus patients treated prior the decision received 2.5mg BI 894999 and patients treated after the decision received 2mg . For Phase Ib - Schedule C NC, the dose was lowered since DMC reclaimed the MTD as 6/3mg on 08Jul2020 after 1 patient already treated with 7/3.5mg, so the first patient in NC and all the following patients were treated with 6/3mg.
Groups:
- Phase Ia - Schedule A: 0.2 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 0.2 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule A: 0.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 0.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule A: 1 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 1 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule A: 1.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 1.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule A: 2 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 2 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule A: 5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
- Phase Ia - Schedule B: 1.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 1.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule B: 2 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 2 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule B: 2.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally 2.5 mg of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule C: 5/2.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 5 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 2.5 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ia - Schedule C: 6/3 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 6 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 3 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ia - Schedule C: 7/3.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 7 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 3.5 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients): Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally 1.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients): Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally 2 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients): Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally 2.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients): Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 4 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 2 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients): Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 5 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 2.5 mg of BI 894999, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients): This arm included adult patients diagnosed with small cell lung cancer (SCLC). SCLC patients were initialy administered 2.5 mg of BI 894999. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
  The Data Monitoring Committee decided on 28 November 2018 to lower the 2.5 mg BI 894999 dose due to safety concerns to 2mg, therefore patients treated before the decision were administered 2.5mg, and patients treated after the decision were administered 2mg.
- Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients): Adult patients diagnosed with colorectal cancer (CRC) were administered orally 2.5 milligram (mg) of BI 894999. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
- Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients): This arm included adult patients diagnosed with metastatic castrate resistant prostate cancer (mCRPC).
  MCRPC patients were initialy administered 2.5 mg of BI 894999. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
  The Data Monitoring Committee decided on 28 November 2018 to lower the 2.5 mg BI 894999 dose due to safety concerns to 2mg, therefore patients treated before the decision were administered 2.5mg, and patients treated after the decision were administered 2mg.
- Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients): Adult patients diagnosed with NUT carcinoma (NC) were administered orally 2.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days. The 2.5 mg dose could be reduced to 2 mg in case of adverse events.
- Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients): This arm included adult patients diagnosed with NUT carcinoma (NC). The DMC reclaimed the maximum tolerated dose (MTD) as 6/3mg on 08 July 2020 after 1 patient was already treated with 7/3.5mg, so the first patient in NC and all the following patients were treated with 6/3mg.
  Patients in were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 6 milligram (mg) of BI 894999, followed by six days intake of the maintenance dose of 3 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C).
Period: Overall Study
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Started | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 8 | 4 | 2 | 2 | 2 | 12 | 14 | 11 | 20 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 8 | 4 | 2 | 2 | 2 | 12 | 14 | 11 | 20 | 22
Not completed — Progressive disease | 2 | 2 | 3 | 5 | 3 | 0 | 5 | 5 | 11 | 3 | 10 | 8 | 8 | 2 | 2 | 2 | 1 | 9 | 12 | 7 | 16 | 18
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Other Adverse Events | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 1
Not completed — Refused to continue trial medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — other reasons than listed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: For Phase Ib - Schedule B SCLC, Phase Ib - Schedule B mCRPC, DMC decided on 28Nov2018 to lower the dose of SCLC and mCRPC due to safety concern, thus patients treated prior the decision received 2.5mg BI 894999 and patients treated after the decision received 2mg . For Phase Ib - Schedule C NC, the dose was lowered since DMC reclaimed the MTD as 6/3mg on 08Jul2020 after 1 patient already treated with 7/3.5mg, so the first patient in NC and all the following patients were treated with 6/3mg.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients) | Total
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 8 | 4 | 2 | 2 | 2 | 12 | 14 | 11 | 20 | 22 | 174
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (10.6) | 69.5 (2.1) | 46.7 (9.3) | 57.5 (11.9) | 53.5 (18.1) | 54.5 (26.2) | 60.7 (10.8) | 61.5 (13.0) | 64.5 (7.5) | 63.3 (12.8) | 59.7 (12.0) | 62.5 (6.5) | 71.4 (10.9) | 78.8 (9.0) | 68.5 (2.1) | 68.5 (2.1) | 79.0 (9.9) | 63.5 (7.3) | 66.2 (6.3) | 69.7 (4.1) | 44.4 (13.9) | 40.5 (16.5) | 58.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 2 | 6 | 0 | 3 | 1 | 4 | 2 | 5 | 7 | 1 | 1 | 1 | 0 | 1 | 5 | 6 | 0 | 5 | 8 | 61
  Male | 1 | 2 | 1 | 4 | 0 | 2 | 3 | 5 | 9 | 2 | 10 | 5 | 7 | 3 | 1 | 2 | 1 | 7 | 8 | 11 | 15 | 14 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 6
  Not Hispanic or Latino | 2 | 2 | 3 | 6 | 5 | 2 | 6 | 6 | 13 | 4 | 14 | 10 | 2 | 4 | 2 | 2 | 1 | 8 | 8 | 9 | 17 | 17 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 4 | 5 | 2 | 3 | 4 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  White | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 2 | 4 | 2 | 1 | 0 | 7 | 9 | 8 | 14 | 16 | 140
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 2 | 4 | 5 | 2 | 3 | 4 | 27

OUTCOME MEASURES:

1. Primary Outcome: Phase Ia: Number of Patients With DLTs Observed in the First Cycle
Description: Number of patients with Dose Limiting Toxicities (DLTs) observed in the first treatment cycle of Phase Ia is reported.
  The following drug related adverse events (AEs) qualified as DLT:
  * any Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 non haematological toxicity considered related to trial medication with the following exceptions:
    * inadequately treated nausea, vomiting or diarrhoea. For fatigue, if present at baseline, there had to be an increase of ≥2 grades
    * electrolytes abnormalities that were corrected within 72 hours with treatment
  * any haematologic AE related to the trial medication defined as follows:
    * CTCAE grade ≥4 neutropenia lasting ≥ 7 days and/or complicated by infection, or
    * CTCAE grade ≥4 thrombocytopenia, or
    * CTCAE grade≥ 3 thrombocytopenia coupled with grade ≥ 2 of bleeding, or
    * febrile neutropenia CTCAE grade 3 or higher.
  * any other drug-related AE preventing the patient from taking his treatment according to the given schedule.
Time Frame: First treatment cycle (the first 21 days for Schedules A and B, the first 28 days for Schedule C).
Population: Maximum Tolerated Dose (MTD) Evaluation Set (MTDS): Included all patients in the treated set (TS) of Phase 1a who were not replaced for the MTD determination.
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ia - Schedule A: 1.5 mg BI 894999: Adult patients with a confirmed diagnosis of advanced, unresectable and/or metastatic malignant solid tumours who had failed conventional treatment or for whom no therapy of proven efficacy existed or who were not amenable to standard therapies were administered 1.5 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule A was a continuous daily intake in cycles of 21 days.
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 6 | 2 | 5 | 6 | 12 | 3 | 12 | 10 | 8 | 3 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 2 | 0 | 2 | 4 | 1 | 1 | 2 | 0 | 0

2. Primary Outcome: Phase Ib: Number of Patients With DLTs Observed During the On-treatment Period
Description: Number of patients with Dose Limiting Toxicities (DLTs) observed during the on-treatment period of Phase Ib is reported.
  The following drug related adverse events (AEs) qualified as DLT:
  * any Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 non haematological toxicity considered related to trial medication with the following exceptions:
    * inadequately treated nausea, vomiting or diarrhoea. For fatigue, if present at baseline, there had to be an increase of ≥2 grades
    * electrolytes abnormalities that were corrected within 72 hours with treatment
  * any haematologic AE related to the trial medication defined as follows:
    * CTCAE grade ≥4 neutropenia lasting ≥ 7 days and/or complicated by infection, or
    * CTCAE grade ≥4 thrombocytopenia, or
    * CTCAE grade≥ 3 thrombocytopenia coupled with grade ≥ 2 of bleeding, or
    * febrile neutropenia CTCAE grade 3 or higher.
  * any other drug-related AE preventing the patient from taking his treatment according to the given schedule.
Time Frame: Date of the first administration of study treatment until date of the last administration of study treatment + 30 days residual effect period, up to 883 days.
Population: For Phase Ib - Schedule B SCLC, Phase Ib - Schedule B mCRPC, DMC decided on 28Nov2018 to lower the dose of SCLC and mCRPC due to safety concern, thus patients treated prior the decision received 2.5mg BI 894999 and patients treated after the decision received 2mg. For Phase Ib - Schedule C NC, the dose was lowered since DMC reclaimed the MTD as 6/3mg on 08Jul2020 after 1 patient already treated with 7/3.5mg, so the first patient in NC and all the following patients were treated with 6/3mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Number analyzed (Participants) | 12 | 14 | 11 | 20 | 22
Participants | 3 | 2 | 7 | 2 | 3

3. Secondary Outcome: Phase Ia: Number of Patients With DLTs Observed During the On-treatment Period
Description: Number of patients with DLTs observed during the on-treatment period of Phase Ia is reported.
  The following drug related adverse events (AEs) qualified as DLT:
  * any Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 non haematological toxicity considered related to trial medication with the following exceptions:
    * inadequately treated nausea, vomiting or diarrhoea. For fatigue, if present at baseline, there had to be an increase of ≥2 grades
    * electrolytes abnormalities that were corrected within 72 hours with treatment
  * any haematologic AE related to the trial medication defined as follows:
    * CTCAE grade ≥4 neutropenia lasting ≥ 7 days and/or complicated by infection, or
    * CTCAE grade ≥4 thrombocytopenia, or
    * CTCAE grade≥ 3 thrombocytopenia coupled with grade ≥ 2 of bleeding, or
    * febrile neutropenia CTCAE grade 3 or higher.
  * any other drug-related AE preventing the patient from taking his treatment according to the given schedule.
Time Frame: Date of the first administration of study treatment until date of the last administration of study treatment + 30 days residual effect period, up to 463 days.
Population: Included all patients in Phase 1a who were dispensed study treatment and were documented to have taken at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 8 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 2 | 4 | 2 | 1 | 0 | 3 | 1 | 3 | 4 | 1 | 2 | 2 | 1 | 2

4. Secondary Outcome: Phase Ia and Phase Ib: Area Under the Concentration-time Curve of BI 894999 in Plasma Over the Time Interval From 0 to 24 Hours After Administration of the First Dose (AUC0-24)
Description: Area under the concentration-time curve of BI 894999 in plasma over the time interval from 0 to 24 hours after administration of the first dose (AUC0-24) for Phase Ia and Phase Ib is reported.
Time Frame: 5 minutes (min) before and at 30 min, 1 hour (h), 2h, 3h, 4h, 6h, 8h and 23h55min after administration of first BI 894999 dose on Day 1 of Cycle 1.
Population: Pharmacokinetic (PK) analysis Set (PKS): Included all patients in the treated set (TS) who have at least one evaluable PK parameters.
  In phase Ib, solid tumor patients (SCLC, mCRPC, CRC and NC) are combined by dose level (2 or 2.5mg) as data of all solid tumor patients were needed since no differences were expected, but the NC patients alone were differentiated in an additional subgroup as it was the initial indication for BI 894999.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole * hour /Liter (nmol*h/L)
Groups:
- Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients): Adult patients diagnosed with NUT carcinoma (NC) were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 7 milligram (mg) of BI 894999, followed by six days intake of the maintenance dose of 3.5 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ib - Schedule B: BI 894999 2 mg (Solid Tumours Including NC): Adult patients diagnosed with one of the following cancer types small cell lung cancer (SCLC); metastatic castrate resistant prostate cancer (mCRPC); NUT carcinoma (NC) were administered orally 2 milligram (mg) of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC): Adult patients diagnosed with one of the following cancer types small cell lung cancer (SCLC); metastatic castrate resistant prostate cancer (mCRPC); colorectal cancer (CRC); NUT carcinoma (NC) were administered orally 2.5 milligram (mg) of BI 894999, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients): Adult patients diagnosed with NUT carcinoma (NC) were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 6 milligram (mg) of BI 894999, followed by six days intake of the maintenance dose of 3 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C).
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) | Phase Ib - Schedule B: BI 894999 2 mg (Solid Tumours Including NC) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 4 | 0 | 3 | 4 | 11 | 4 | 15 | 12 | 7 | 4 | 2 | 2 | 0 | 1 | 9 | 17 | 42 | 2
nanomole * hour /Liter (nmol*h/L) | 4.36 (21.1) | 6.43 (2.78) | 20.5 (16.8) | 34.0 (69.4) | 64.9 (71.0) |  | 27.7 (81.5) | 44.8 (34.8) | 51.5 (41.7) | 123 (37.6) | 212 (45.5) | 230 (27.3) | 31.7 (33.4) | 48.0 (26.9) | 53.3 (6.91) | 138 (7.52) |  | NA (NA) — AUC0-24 could not be provided to reduce the risk of patient re-identificaton. | 39.2 (38.8) | 56.9 (58.6) | 67.6 (50.9) | 214 (6.01)

5. Secondary Outcome: Phase Ia and Phase Ib: Maximum Measured Concentration of BI 894999 in Plasma After the First Dose (Cmax)
Description: Maximum measured concentration of BI 894999 in plasma after the first dose (Cmax) for Phase 1a and Phase 1b is reported.
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) analysis Set (PKS): Included all patients in the treated set (TS) who have at least one evaluable PK parameters.
  In phase Ib, solid tumor patients (SCLC, mCRPC, CRC and NC) are combined by dose level (2 or 2.5mg) as data of all solid tumor patients were needed since no differences were expected, but the NC patients alone were differentiated in an additional subgroup as it was the initial indication for BI894999.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/L (nmol/L)
Groups:
- Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients): Adult patients diagnosed with NUT carcinoma (NC) who were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 7 milligram (mg) of BI 894999, followed by six days intake of the maintenance dose of 3.5 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) | Phase Ib - Schedule B: BI 894999 2 mg (Solid Tumours Including NC) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 4 | 2 | 3 | 4 | 11 | 4 | 15 | 12 | 7 | 4 | 2 | 2 | 1 | 1 | 9 | 17 | 44 | 15
nanomole/L (nmol/L) | 0.393 (35.6) | 0.569 (46.2) | 1.75 (31.6) | 3.79 (84.0) | 7.39 (56.0) | 16.2 (68.0) | 3.00 (155) | 3.93 (50.2) | 4.48 (46.6) | 12.0 (85.1) | 19.4 (58.4) | 21.0 (48.3) | 2.98 (34.9) | 4.49 (36.0) | 4.75 (0.595) | 13.9 (12.8) | NA (NA) — Cmax could not be provided to reduce the risk of patient re-identificaton. | NA (NA) — Cmax could not be provided to reduce the risk of patient re-identificaton. | 4.10 (37.8) | 4.88 (50.1) | 6.01 (59.6) | 18.8 (55.8)

6. Secondary Outcome: Phase Ia and Phase Ib: Area Under the Concentration-time Curve of BI 894999 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ, ss)
Description: Area under the concentration-time curve of BI 894999 in plasma at steady state over a uniform dosing interval τ (AUCτ, ss) for Phase Ia and Ib is reported. The dosing interval is 24 hours (h) for all dose groups.
Time Frame: 5 minutes (min) before and at 30 min, 1 hour (h), 2h, 3h, 4h, 6h, 8h, and at 23h55min (Schedule A) or 24h (Schedule B & C) following administration on day 14 (Schedule A & B) or day 21 (Schedule C).
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole *hour/Liter (nmol*h/)L
Groups:
- Phase Ib - Schedule B: 2 mg BI 894999 (NC Patients Only): Adult patients diagnosed with NUT carcinoma (NC) who were administered during the first cycle 2.5 milligram (mg) BI 894999 according to Schedule B and then the dosage was decreased at steady state to 2 mg of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC): Adult patients diagnosed with one of the following cancer types small cell lung cancer (SCLC); metastatic castrate resistant prostate cancer (mCRPC); colorectal cancer (CRC); NUT carcinoma (NC) who were administered orally 2.5 milligram (mg) of BI 894999, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) | Phase Ib - Schedule B: 2 mg BI 894999 (NC Patients Only) | Phase Ib - Schedule B: BI 894999 2 mg (Solid Tumours Including NC) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 4 | 4 | 1 | 4 | 6 | 11 | 3 | 14 | 5 | 6 | 3 | 1 | 1 | 1 | 0 | 1 | 10 | 14 | 33 | 11
nanomole *hour/Liter (nmol*h/)L | 10.3 (72.6) | 17.9 (46.4) | 54.6 (40.4) | 76.4 (26.6) | 119 (90.3) | NA (NA) — AUCτ, ss could not be provided to reduce the risk of patient re-identificaton. | 62.6 (49.2) | 81.1 (32.1) | 87.0 (28.3) | 144 (46.4) | 176 (37.0) | 226 (63.2) | 70.3 (38.5) | 120 (19.6) | NA (NA) — AUCτ, ss could not be provided to reduce the risk of patient re-identificaton. | NA (NA) — AUCτ, ss could not be provided to reduce the risk of patient re-identificaton. | NA (NA) — AUCτ, ss could not be provided to reduce the risk of patient re-identificaton. |  | NA (NA) — AUCτ, ss could not be provided to reduce the risk of patient re-identificaton. | 73.6 (58.2) | 94.9 (43.9) | 125 (50.4) | 149 (56.7)

7. Secondary Outcome: Phase Ia and Phase Ib: Maximum Measured Concentration of BI 894999 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax, ss)
Description: Maximum measured concentration of BI 894999 in plasma at steady state over a uniform dosing interval τ (Cmax, ss) for Phase Ia and Phase Ib is reported. The dosing interval is 24 hours (h) for all dose groups.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Groups:
- Phase Ib - Schedule B: 2 mg BI 894999 (NC Patients Only): Adult patients diagnosed with NUT carcinoma (NC) were administered during the first cycle 2.5 milligram (mg) BI 894999 according to Schedule B and then the dosage was decreased at steady state to 2 mg of BI 894999 once daily, in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water. Schedule B was a continuous intake for 14 days followed by one week off treatment in cycles of 21 days.
- Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients): Adult patients diagnosed with NUT carcinoma (NC) who were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 6 milligram (mg) of BI 894999, followed by six days intake of the maintenance dose of 3 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C).
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) | Phase Ib - Schedule B: 2 mg BI 894999 (NC Patients Only) | Phase Ib - Schedule B: BI 894999 2 mg (Solid Tumours Including NC) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule B: BI 894999 2.5 mg (Solid Tumours Including NC) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 6 | 1 | 4 | 6 | 11 | 3 | 14 | 5 | 6 | 3 | 1 | 1 | 1 | 0 | 1 | 10 | 14 | 33 | 11
nanomole/Liter (nmol/L) | 0.697 (59.8) | 1.26 (24.9) | 4.06 (61.7) | 5.25 (60.1) | 11.6 (54.4) | NA (NA) — Cmax, ss could not be provided to reduce the risk of patient re-identificaton. | 4.75 (46.9) | 5.62 (27.7) | 6.94 (42.0) | 11.4 (56.1) | 13.1 (41.8) | 17.1 (63.6) | 5.48 (32.7) | 7.67 (8.44) | NA (NA) — Cmax, ss could not be provided to reduce the risk of patient re-identificaton. | NA (NA) — Cmax, ss could not be provided to reduce the risk of patient re-identificaton. | NA (NA) — Cmax, ss could not be provided to reduce the risk of patient re-identificaton. |  | NA (NA) — Cmax, ss could not be provided to reduce the risk of patient re-identificaton. | 6.51 (70.0) | 7.68 (45.4) | 10.4 (59.4) | 11.2 (60.1)

8. Secondary Outcome: Phase Ia and Phase Ib: Objective Response (OR)
Description: OR was defined as best overall response (BOR) of complete response (CR) or partial response (PR) with tumour assessment during treatment period for each schedule.
  For DLBCL patients, a minor response according to Response Evaluation Criteria In Lymphoma 2017 (RECIL 2017) was not part of an objective response.
  BOR was determined from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent, according to the following criteria depending on the type of cancer:
  * solid tumour patients and mCRPC patients with measurable disease: CT and/ or MRI according to RECIST v1.1, every 2 cycles;
  * mCRPC patients without measurable disease: bone scan and PSA level according to Prostate Cancer Clinical Trials Working Group 3, every 4 cycles;
  * DLBCL patients:FDG-PET/CT scans according to RECIL 2017; every 2 cycles.
Time Frame: Up to 15 months for Phase 1a and up to 28 months for Phase Ib.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 6 | 2 | 6 | 6 | 13 | 4 | 15 | 12 | 8 | 4 | 2 | 2 | 2 | 12 | 14 | 11 | 20 | 22
Participants | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2

9. Secondary Outcome: Phase Ib: Progression-free Survival or (PFS) or Radiological PFS for mCRPC Patients With Non-measurable Disease by RECIST v1.1
Description: Progression-free survival (PFS) was defined as the time from date of start of BI 894999 to the date of objective disease progression ((PD) defined as 20% increase in the sum of the longest diameter of target lesions) or death, whichever is earlier for SCLC patients, CRC patients, mCRPC patients with measurable disease by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and NC patients, with tumour assessment every 2 cycles according to RECIST v1.1 during treatment period or Radiological PFS with tumour assessment by bone scan every 4 cycles for mCRPC patients with non-measurable disease by RECIST v1.1.
  For patients with 'event' as an outcome for PFS:
  - PFS [days] = date of outcome - date of first treatment administration + 1.
  For patients with 'censored' as an outcome for PFS:
  - PFS (censored) [days] = date of outcome - date of first treatment administration + 1.
  The Kaplan-Meier method was used to calculate the estimates.
Time Frame: Up to 28 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Number analyzed (Participants) | 12 | 14 | 11 | 20 | 22
Weeks | 5.6 [5.3 to 6.1] | 5.6 [4.4 to 10.7] | 11.9 [8.1 to 24.4] | 6.9 [6.0 to 11.1] | 7.8 [4.0 to 13.0]

10. Secondary Outcome: Phase Ib: Best Overall Response
Description: Best overall response (BOR) was determined from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent, according to the following criteria depending on the type of cancer:
  * solid tumour patients and mCRPC patients with measurable disease: Computerized tomography (CT) and/ or magnetic resonance imaging (MRI) according to RECIST v1.1, every 2 cycles;
  * mCRPC patients without measurable disease: bone scan and PSA level according to Prostate Cancer Clinical Trials Working Group 3, every 4 cycles.
Time Frame: Imaging and assessment performed every 2 cycles (solid tumours patients) or 4 cycles (mCRPC patients) for the entire treatment period, up to 28 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Number analyzed (Participants) | 12 | 14 | 11 | 20 | 22
Participants
  Complete response | 0 | 0 | 0 | 0 | 1
  Partial response | 0 | 0 | 1 | 1 | 1
  Stable disease | 1 | 2 | 2 | 7 | 6
  Progressive disease | 8 | 10 | 4 | 9 | 9
  Not evaluable | 3 | 2 | 4 | 3 | 5
  Not assessed | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Phase Ib: Overall Survival
Description: Overall survival (OS) was defined as the time from first administration of BI 894999 until death from any cause in patients with NUT carcinoma.
  For patients with 'event' as an outcome for OS:
  - OS [days] = date of outcome - date of first treatment administration + 1.
  For patients with 'censored' as an outcome for OS:
  - OS (censored) [days] = date of outcome - date of first treatment administration + 1.
  The Kaplan-Meier method was used to calculate the estimates.
Time Frame: Up to 28 months.
Population: Patients in NC Schedules B and C in Phase Ib dose expansion and after approval of protocol version 11.0 and gave consent to the collection of overall survival status.
  For "Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC patients)" arm, the dose was lowered since DMC reclaimed the MTD as 6/3mg on 08Jul2020 after 1 patient already treated with 7/3.5mg, so the first patient in NC and all the following patients were treated with 6/3mg.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: 6/3 or 7/3.5 mg BI 894999 (NC Patients)
Number analyzed (Participants) | 1 | 22
Weeks | 6.6 [NA to NA] — 95% Confidence Interval could not be calculated due to insufficient number of participants with events. | 15.4 [7.6 to 32.3]

12. Secondary Outcome: Phase Ib: Prostate Specific Antigen (PSA) Response in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Description: PSA response was defined as a decline in PSA value ≥50% from baseline (which is confirmed by a second value 3 to 4 weeks apart).
Time Frame: Up to 93 days.
Population: mCRPC Schedule B in Phase Ib dose expansion (mCRPC): Included all mCRPC patients in the treated set who were treated in Phase Ib with Schedule B.
  For "Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC patients)", DMC decided on 28Nov2018 to lower the dose of mCRPC due to safety concern, thus patients treated prior the decision received 2.5mg BI 894999 and patients treated after the decision received 2mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib - Schedule B: 2 or 2.5 mg BI 894999 (mCRPC Patients)
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: [All-Cause Mortality]: From first date of dosing until end of study, up to 1309 days for Phase Ia and up to 860 days for Phase Ib. [Serious and Other Adverse Events]: From first date of dosing of study treatment until date of the last dosing of study treatment + 30 days residual effect period, up to 463 days for Phase 1a and up to 883 days for Phase Ib.
Description: Treated Set (TS): Included all patients who were dispensed study treatment and were documented to have taken at least one dose of the study treatment.
Groups:
- Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients: Adult patients with histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) were administered orally once daily on Day 1 and on Day 15 of each cycle a loading dose of 4 milligram (mg) of BI 894999, followed by six days daily intake of the maintenance dose of 2 mg of BI 894999 once daily, followed by one week off, repeated every two weeks in cycles of 28 days (Schedule C). The loading and the maintenance dose were administered in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water.
- Phase Ib - Schedule B: 2.5 mg BI 894999 (SCLC Patients): Adult patients diagnosed with small cell lung cancer (SCLC) were administered 2.5 milligram (mg) of BI 894999 once daily. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
- Phase Ib - Schedule B: 2 mg BI 894999 (SCLC Patients): Adult patients diagnosed with small cell lung cancer (SCLC) were administered orally 2 milligram (mg) of BI 894999 once daily. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
- Phase Ib - Schedule B: 2.5 mg BI 894999 (mCRPC Patients): Adult patients diagnosed with metastatic castrate resistant prostate cancer (mCRPC) were administered orally 2.5 milligram (mg) of BI 894999 once daily. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
- Phase Ib - Schedule B: 2 mg BI 894999 (mCRPC Patients): Adult patients diagnosed with metastatic castrate resistant prostate cancer (mCRPC) were administered orally 2 milligram (mg) of BI 894999 once daily. BI 894999 administration was performed in the morning, after an overnight fast, 1 hour before breakfast with at least 250 milliliter (mL) of water according to Schedule B (continuous intake for 14 days followed by one week off treatment in cycles of 21 days).
Arm/Group | Phase Ia - Schedule A: 0.2 mg BI 894999 | Phase Ia - Schedule A: 0.5 mg BI 894999 | Phase Ia - Schedule A: 1 mg BI 894999 | Phase Ia - Schedule A: 1.5 mg BI 894999 | Phase Ia - Schedule A: 2 mg BI 894999 | Phase Ia - Schedule A: 5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 | Phase Ia - Schedule B: 2 mg BI 894999 | Phase Ia - Schedule B: 2.5 mg BI 894999 | Phase Ia - Schedule C: 5/2.5 mg BI 894999 | Phase Ia - Schedule C: 6/3 mg BI 894999 | Phase Ia - Schedule C: 7/3.5 mg BI 894999 | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2 mg BI 894999 (SCLC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2 mg BI 894999 (mCRPC Patients) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 1/6 | 1/6 | 0/2 | 1/6 | 1/6 | 2/13 | 0/4 | 2/15 | 1/12 | 0/8 | 0/4 | 0/2 | 1/2 | 0/2 | 0/3 | 1/9 | 0/14 | 0/10 | 0/1 | 5/20 | 2/21 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 0/3 | 3/6 | 2/6 | 1/2 | 3/6 | 3/6 | 6/13 | 2/4 | 8/15 | 8/12 | 3/8 | 2/4 | 2/2 | 1/2 | 0/2 | 2/3 | 3/9 | 8/14 | 8/10 | 1/1 | 15/20 | 12/21 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 3/3 | 6/6 | 6/6 | 2/2 | 6/6 | 6/6 | 12/13 | 4/4 | 15/15 | 12/12 | 8/8 | 4/4 | 2/2 | 2/2 | 2/2 | 3/3 | 9/9 | 14/14 | 10/10 | 1/1 | 20/20 | 21/21 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia - Schedule A: 0.2 mg BI 894999 (N=2) | Phase Ia - Schedule A: 0.5 mg BI 894999 (N=2) | Phase Ia - Schedule A: 1 mg BI 894999 (N=3) | Phase Ia - Schedule A: 1.5 mg BI 894999 (N=6) | Phase Ia - Schedule A: 2 mg BI 894999 (N=6) | Phase Ia - Schedule A: 5 mg BI 894999 (N=2) | Phase Ia - Schedule B: 1.5 mg BI 894999 (N=6) | Phase Ia - Schedule B: 2 mg BI 894999 (N=6) | Phase Ia - Schedule B: 2.5 mg BI 894999 (N=13) | Phase Ia - Schedule C: 5/2.5 mg BI 894999 (N=4) | Phase Ia - Schedule C: 6/3 mg BI 894999 (N=15) | Phase Ia - Schedule C: 7/3.5 mg BI 894999 (N=12) | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) (N=8) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) (N=4) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) (N=2) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients (N=2) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) (N=2) | Phase Ib - Schedule B: 2.5 mg BI 894999 (SCLC Patients) (N=3) | Phase Ib - Schedule B: 2 mg BI 894999 (SCLC Patients) (N=9) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) (N=14) | Phase Ib - Schedule B: 2.5 mg BI 894999 (mCRPC Patients) (N=10) | Phase Ib - Schedule B: 2 mg BI 894999 (mCRPC Patients) (N=1) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) (N=20) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients) (N=21) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Euthanasia (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jugular vein distension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia - Schedule A: 0.2 mg BI 894999 (N=2) | Phase Ia - Schedule A: 0.5 mg BI 894999 (N=2) | Phase Ia - Schedule A: 1 mg BI 894999 (N=3) | Phase Ia - Schedule A: 1.5 mg BI 894999 (N=6) | Phase Ia - Schedule A: 2 mg BI 894999 (N=6) | Phase Ia - Schedule A: 5 mg BI 894999 (N=2) | Phase Ia - Schedule B: 1.5 mg BI 894999 (N=6) | Phase Ia - Schedule B: 2 mg BI 894999 (N=6) | Phase Ia - Schedule B: 2.5 mg BI 894999 (N=13) | Phase Ia - Schedule C: 5/2.5 mg BI 894999 (N=4) | Phase Ia - Schedule C: 6/3 mg BI 894999 (N=15) | Phase Ia - Schedule C: 7/3.5 mg BI 894999 (N=12) | Phase Ia - Schedule B: 1.5 mg BI 894999 (DLBCL Patients) (N=8) | Phase Ia - Schedule B: 2 mg BI 894999 (DLBCL Patients) (N=4) | Phase Ia - Schedule B: 2.5 mg BI 894999 (DLBCL Patients) (N=2) | Phase Ia - Schedule C: 4/2 mg BI 894999 (DLBCL Patients (N=2) | Phase Ia - Schedule C: BI 894999 5/2.5 mg (DLBCL Patients) (N=2) | Phase Ib - Schedule B: 2.5 mg BI 894999 (SCLC Patients) (N=3) | Phase Ib - Schedule B: 2 mg BI 894999 (SCLC Patients) (N=9) | Phase Ib - Schedule B: 2.5 mg BI 894999 (CRC Patients) (N=14) | Phase Ib - Schedule B: 2.5 mg BI 894999 (mCRPC Patients) (N=10) | Phase Ib - Schedule B: 2 mg BI 894999 (mCRPC Patients) (N=1) | Phase Ib - Schedule B: 2.5 mg BI 894999 (NC Patients) (N=20) | Phase Ib - Schedule C: BI 894999 6/3 mg (NC Patients) (N=21) | Phase Ib - Schedule C: BI 894999 7/3.5 mg (NC Patients) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 4 | 0 | 5 | 6 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 9 | 1 | 11 | 6 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 5 | 1 | 0 | 3 | 6 | 2 | 8 | 7 | 4 | 4 | 2 | 0 | 1 | 2 | 2 | 5 | 5 | 0 | 5 | 5 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 2 | 6 | 3 | 8 | 3 | 2 | 3 | 2 | 2 | 2 | 0 | 3 | 8 | 6 | 0 | 4 | 9 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 4 | 2 | 2 | 1 | 4 | 6 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 6 | 5 | 0 | 4 | 4 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 1 | 3 | 4 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 6 | 0 | 1 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 3 | 4 | 4 | 2 | 1 | 3 | 6 | 2 | 8 | 10 | 0 | 3 | 1 | 1 | 0 | 1 | 3 | 6 | 6 | 0 | 8 | 10 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 5 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iodine allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Activated partial thromboplastin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 6 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Blood antidiuretic hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cortisol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Echocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 8 | 8 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 3 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 4 | 1 | 4 | 6 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 7 | 6 | 1 | 5 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 8 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agnosia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 4 | 0 | 4 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 2 | 5 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 3 | 4 | 0 | 3 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This trial was closed in accordance with protocol-defined criteria for stopping the trial following assessments of futility. Trial was completed as described in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02516553/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02516553/SAP_001.pdf